CLINICAL TRIAL: NCT01686165
Title: A Phase II Exploratory Study of PXD-101(Belinostat) Followed by Zevalin in Patients With Relapsed Aggressive High-Risk Lymphoma
Brief Title: Belinostat and Yttrium Y 90 Ibritumomab Tiuxetan in Patients W/Relapsed Aggressive B-Cell NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0288-04; NCI-2012-01131 (Other: CTRP (Clinical Trial Reporting Program)); 1200000288 (Other: UofA IRB #); P30CA023074 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Anaplastic Large Cell Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — belinostat; Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belinostat Yttrium Ibritumomab Tiuxetan (Experimental): Patients receive belinostat IV over 30-60 minutes on days 1-5. Treatment with belinostat repeats every 21 days for 2 courses. Patients then receive rituximab IV on days 1 and either 7, 8, or 9, and yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 50. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: belinostat; Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Drug: belinostat — Given IV
  Other Names: PXD101
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Radiation: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan

SUMMARY:
This study looks at what effects (good and bad) a drug called PXD-101 (belinostat) in combination with the radioactive drug Zevalin (yttrium Y 90 ibritumomab tiuxetan) has on patients with relapsed aggressive (high-risk) non-Hodgkin lymphoma. Studies in the laboratory suggest that drugs such as PXD101 can act upon specific cancer cell processes to cause either death of the cancer cells or prevention of their growth. In human studies with a small number of patients with this lymphoma, PXD-101 has shown the ability to shrink and slow tumor growth. When Zevalin is delivered directly to the tumor, the lymphoma cells are destroyed and this may result in the disappearance of the tumor (remission)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To document the complete response rate and overall response for patients with relapsed aggressive high-risk non-Hodgkin's lymphoma treated with two cycles PXD-101 followed by one cycle of Zevalin.

SECONDARY OBJECTIVES:

I. To estimate 2-year progression-free survival in patients with relapsed aggressive high-risk non-Hodgkin's lymphoma treated with two cycles PXD-101 followed by one cycle of Zevalin.

II. To evaluate the toxicity of two cycles PXD-101 and one cycle of Zevalin in patients with relapsed aggressive high-risk non-Hodgkin's lymphoma.

OUTLINE:

Patients receive belinostat intravenously (IV) over 30-60 minutes on days 1-5. Treatment with belinostat repeats every 21 days for 2 courses. Patients then receive rituximab IV on days 1 and either 7, 8, or 9, and yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 50. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed, CD20 positive diffuse large B-cell lymphoma, primary mediastinal b-cell lymphoma, mantel cell lymphoma, transformed indolent lymphoma, high grade-B-cell lymphoma; AND bone marrow must show =< 20% CD20+ B-cells with >= 15% cellularity within 42 days of study registration
* Any stage disease
* Patients must have been previously treated:

  * >= 3rd line if bone marrow transplant (BMT) candidate OR
  * >= 2nd line if not BMT candidate OR
  * >= 2nd relapse for BMT candidate OR
  * >= 1st relapse for non- BMT candidate
* Must have a diagnostic quality CT scan of the chest, abdomen and pelvis OR baseline PET-CT scan performed within 28 days prior to registration
* Must have bidimensionally measurable disease with lesions at least 1.5 cm in one dimension ALL measurable disease must be assessed within 28 days of registration
* To determine prior drug regimens: radiation therapy counts as 1 treatment, BMT including induction counts as one treatment, radioimmunotherapy is not considered a chemotherapy regimen, rituximab alone is not considered a treatment; all prior therapy must have been completed at least 30 days prior to registration; patients should not have taken valproic acid, or any other histone deacetylase inhibitor (eg., vorinostat, romidepsin), for at least 30 days prior to registration; patients must have recovered from any toxicities related to therapies prior to registration
* No clinical evidence of CNS involvement by lymphoma, any lab (eg., LDH or radiographic tests performed to access CNS involvement must be negative and must be performed within 42 days prior to registration
* Unilateral or bilateral bone marrow biopsy performed within 42 days prior to registration
* Life expectancy of greater than 3 months
* Karnofsky performance status >= 60%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* AST (SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Total bilirubin =< 1.5 X institutional upper limit of normal (unless associated with Gilbert's syndrome)
* Serum creatinine < 2 x institutional upper limit of normal OR
* Measured creatinine clearance >= 60 mL/min
* LDH < 1.50 X institutional upper limit of normal
* EKG with no significant abnormalities within 28 days prior to registration
* Women of child-bearing potential and men must agree to use adequate contraception

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 30 days (6 weeks for nitrosoureas or mitomycin C) prior to study screening or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Prior radioimmunotherapy
* Pregnant or nursing
* Clinical evidence of CNS involvement by lymphoma
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PXD-101 or Zevalin or other agents used in the study
* Concomitant medication that may cause Torsade de Pointes, i.e. prolongation of the QT interval > 500 msec
* Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, congestive heart failure related to primary cardiac disease, any condition requiring anti-arrhythmic therapy, ischemic or valvular heart disease, or a myocardial infarction within the past 6 months
* Current long QT syndrome or baseline prolongation of QT/QTcF interval, i.e. demonstration of a QTcF interval > 450 msec
* Clinical evidence of severe peripheral vascular disease, diabetic ulcers or venous stasis ulcers, or history of deep venous or arterial thrombosis within 3 months prior to screening
* Known to be human immunodeficiency virus (HIV) positive or with known acquired immunodeficiency syndrome (AIDS) syndrome
* Patients may not be receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O. Persky, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

REFERENCES:
- [Derived] Puvvada SD, Guillen-Rodriguez JM, Rivera XI, Heard K, Inclan L, Schmelz M, Schatz JH, Persky DO. A Phase II Exploratory Study of PXD-101 (Belinostat) Followed by Zevalin in Patients with Relapsed Aggressive High-Risk Lymphoma. Oncology. 2017;93(6):401-405. doi: 10.1159/000479230. Epub 2017 Sep 5. PMID 28869931

RESULTS

PARTICIPANT FLOW:
Groups:
- PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle: Treatment with PXD101 will be administered intravenously** at a dose of 1,000 mg/m2 IV days 1-5 every 21 days for 2 cycles. Yttrium-90 ibritumomab tiuxetan (Zevalin®) Administration. Y-90 Zevalin will be administered to all subjects in accordance with the approved Zevalin product labeling. Treatment will be administered on an outpatient basis.
Period: Overall Study
Arm/Group | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: To document the complete response rate for patients with relapsed aggressive high-risk non-Hodgkin's lymphoma (NHL) treated with two cycles PXD-101 followed by one cycle of the Zevalin regimen.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Overall Response
Description: To document the overall response for patients with relapsed aggressive high-risk non-Hodgkin's lymphoma (NHL) treated with two cycles PXD-101 followed by one cycle of the Zevalin regimen.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Progression-free Survival
Description: Will be estimated using a Kaplan-Meier estimate. The observed 2-year progression-free survival rate will be estimated (with a 95% confidence interval) from the Kaplan-Meier curve.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Occurrence of Adverse Events and Serious Adverse Events
Description: The proportion of patients with a given adverse event will be tabulated and the 95% confidence interval computed.
Time Frame: Up to 30 days after patient receives last dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Three years, six months.
Arm/Group | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle (N=5)
Deep Venous Thrombosis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PXD-101 (d1-d5) for 2 Cycles > Zevalin 1 Cycle (N=5)
Nausea/Vomiting (Gastrointestinal disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Pain (General disorders) | 3
Edema - lower extremity (Vascular disorders) | 2
Increased Serum Creatinine (Blood and lymphatic system disorders) | 2
Sensory Neuropathy (Nervous system disorders) | 2
Hypoglycemia (Endocrine disorders) | 1
Blurred Vision (Eye disorders) | 1
Dizziness (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 1
Otitis Media (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Transaminitis (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes